CLINICAL TRIAL: NCT02169141
Title: Pharmacokinetics of Levofloxacin and Capreomycin in MDR-TB Patients
Brief Title: Pharmacokinetics of Levofloxacin and Capreomycin in Multidrug-Resistant Tuberculosis Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Republican Scientific and Practical Centre for Pulmonology and TB (Unknown); National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Principal Investigator, JWC Alffenaar, PhD PharmD Clinical Pharmacologist Associate Professor, University Medical Center Groningen
Other Study IDs: LC-20
Record Dates: First submitted 2014-06-12; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Tuberculosis
Keywords: pharmacokinetics; pharmacodynamics; MDR-TB; Levofloxacin; Capreomycin
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — Pharmacokinetics

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PK of Levofloxacin-Capreomycin: Pharmacokinetics (PK) in M/XDR-TB patients receiving at least Levofloxacin and Capreomycin as part of their WHO treatment for M/XDR-TB
  Interventions: Other: Pharmacokinetics

INTERVENTIONS:
Other: Pharmacokinetics — multiple blood samples are obtained by means of an indwelling intravenous catheter for calculating PK parameters

SUMMARY:
This is an open label observational pharmacokinetic drug study to evaluate Levofloxacine and Capreomycin in patients with Multidrug-Resistant Tuberculosis (MDR-TB).

DETAILED DESCRIPTION:
Patients receive MDR-TB treatment with o.a. Levofloxacin and Capreomycin. At least one week after start of treatment, the PK samples samples will be obtained via an intravenous catheter at 0, 1, 2, 3, 4, 7, and 12 hours after intake.

ELIGIBILITY:
Inclusion Criteria:

* age> 18yrs
* culture positive
* diagnosis of MDR-TB

Exclusion Criteria:

* DM2
* Pregnancy
* allergy to IV canula material
* insertion of IV canula not possibele

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDR-TB patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
AUC/MIC ratio of Levofloxacin | after day 8 of treatment
  The primary outcome parameter is the ratio of the in vitro minimum inhibitory concentration (MIC) to the area under the serum concentration-time curve (AUC) over 24 hours (AUC0-24h ), [AUC0-24h /MIC], after administration of Levofloxacin.
Cmax/MIC ratio of Capreomycin | after day 8 of treatment
  The primary outcome parameter is the ratio of the in vitro minimum inhibitory concentration (MIC) to the maximum serum concentration, [Cmax/MIC], after administration of Capreomycin.

SECONDARY OUTCOMES:
Volume of Distribution | after day 8 of treatment
  Based on the measured drug concentration during the dosing interval and patient characteristics (height, bodyweight and age) the volume of distribution will be calculated
Clearance | after day 8 of treatment
  Based on the drug concetrations during the dosing interval and patient characteristics (height, bodyweight, age) the drug clearance will be calculated

OTHER OUTCOMES:
PK-model | after day 8 of treatment
  A population PK model will be developed using an iterative 2-stage Bayesian procedure.
Limited sampling strategy | after day 8 of treatment
  Limited sampling strategies were investigated subsequently using a Bayesian analysis. The best possible strategies for will be evaluated by a Bland-Altman analysis for correlation of predicted and observed AUC0-24.

CONTACTS AND LOCATIONS:
Overall Officials: JW C Alffenaar, PhD PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Republican Scientific and Practical Center for TB and Pulmonology, Minsk, Belarus

REFERENCES:
- [Derived] Van't Boveneind-Vrubleuskaya N, Seuruk T, van Hateren K, van der Laan T, Kosterink JGW, van der Werf TS, van Soolingen D, van den Hof S, Skrahina A, Alffenaar JC. Pharmacokinetics of Levofloxacin in Multidrug- and Extensively Drug-Resistant Tuberculosis Patients. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00343-17. doi: 10.1128/AAC.00343-17. Print 2017 Aug. PMID 28507117
- [Derived] Velasquez AMA, Ribeiro WC, Venn V, Castelli S, Camargo MS, de Assis RP, de Souza RA, Ribeiro AR, Passalacqua TG, da Rosa JA, Baviera AM, Mauro AE, Desideri A, Almeida-Amaral EE, Graminha MAS. Efficacy of a Binuclear Cyclopalladated Compound Therapy for Cutaneous Leishmaniasis in the Murine Model of Infection with Leishmania amazonensis and Its Inhibitory Effect on Topoisomerase 1B. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00688-17. doi: 10.1128/AAC.00688-17. Print 2017 Aug. PMID 28507113